CLINICAL TRIAL: NCT05170009
Title: Randomized Double-blind, Placebo-controlled Single Center Pilot Study to Evaluate the Efficacy and Safety of Baloxavir in Combination With Oseltamivir in Adult Allogeneic Bone Marrow Transplant Recipients With Influenza
Brief Title: Baloxavir in Combination With Oseltamivir in Allogenic Bone Marrow Transplant Recipients With Influenza
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Slow enrollment rate
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-12023076
Record Dates: First submitted 2021-12-09; First posted 2021-12-27 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Influenza
Keywords: Influenza; Bone marrow transplant; Flu; Baloxavir Marboxil; Xofluza; Oseltamivir
MeSH Terms: conditions — Influenza, Human | interventions — baloxavir; Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active and standard of care (Active Comparator): Active Baloxavir Marboxil and standard of care Oseltamivir
  Interventions: Drug: Baloxavir Marboxil; Drug: Oseltamivir
- Placebo and standard of care (Placebo Comparator): Placebo-matched Baloxavir Marboxil and standard of care Oseltamivir
  Interventions: Drug: Placebo; Drug: Oseltamivir

INTERVENTIONS:
Drug: Baloxavir Marboxil — Weight-adjusted Baloxavir Marboxil (40 mg for patients weighing <80 kg and 80 mg for those weighing ≥80 kg) at baseline, day 4, and day 7.
  Other Names: Xofluza
  Arms: Active and standard of care
Drug: Placebo — Placebo at baseline, day 4, and day 7.
  Arms: Placebo and standard of care
Drug: Oseltamivir — Oseltamivir 75 mg twice daily for 10 days.
  Other Names: Tamiflu

SUMMARY:
This is a randomized, double-blind, placebo-controlled pilot study of the efficacy and safety of baloxavir in combination with oseltamivir (standard of care) for the treatment of influenza in allogeneic stem cell transplant patients. Although there are no data about this treatment option currently available, the investigator hypothesizes that combination therapy may be more effective in clearing influenza virus infection and decreasing the rate of emergence of resistant influenza in immunocompromised human hosts.

DETAILED DESCRIPTION:
This is a randomized double-blind placebo-controlled pilot study of the efficacy and safety of baloxavir in combination with oseltamivir (standard of care) for the treatment of influenza in allogeneic stem cell transplant patients. 30 SCT recipients will take part in the study. Participants with be randomly assigned (1:1) to either baloxavir + oseltamivir or baloxavir-matched placebo +oseltamivir. Before randomization, patients will be stratified by hospitalization status and influenza type A (yes/no).

Patients in the baloxavir combination arm will receive weight-adjusted baloxavir (40 mg for patients weighing <80 kg and 80 mg for those weighing ≥80 kg) at baseline and at day 4 and day 7. They will also receive oseltamivir 75 mg twice daily for 10 days. Patients in the baloxavir-matched placebo + oseltamivir arm will receive baloxavir-matched placebo at baseline and at day 3 and day 7and oseltamivir 75 mg twice daily for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients: Signed informed consent by any patient capable of giving consent, or, where the patient is not capable of giving consent, by his or her legal/authorized representative
* Age greater than or equal to 18 years at the time of signing the Informed Consent Form/Assent Form
* Ability to comply with the study protocol, in the investigator's judgment
* Have received allogeneic bone marrow transplant
* Tested positive for influenza infection after the onset of symptoms using a polymerase chain reaction (PCR)-based diagnostic assay.
* Presence of (a) fever (≥38.0 °C per tympanic or rectal thermometer; ≥ 37.5 °C per axillary, oral or forehead/temporal thermometer) or (b) any influenza symptoms (cough, sore throat, nasal congestion, headache, feverishness or chills, muscle or joint pain, fatigue).
* The time interval between the diagnosis of influenza and the pre-dose examinations is 48 hours or less.
* For women of childbearing potential: Agreement to remain abstinent (refrain from heterosexual intercourse):
* Women must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 28 days after the last dose of study treatment. Hormonal contraceptive methods must be supplemented by a barrier method. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state greater than or equal to 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

* Patients who have received more than 48 hours of antiviral treatment for the current influenza infection prior to screening
* Patients who have received Baloxavir for the current influenza infection
* Known contraindication to neuraminidase inhibitors
* Patients weighing < 40 kg
* Patients unable to swallow tablets
* Patients with known severe renal impairment (estimated glomerular filtration rate < 30 mL/min/1.73 m2) or receiving continuous renal replacement therapy, hemodialysis, peritoneal dialysis
* Patients with any of the following laboratory abnormalities detected within 24 hours prior to or during screening (according to local laboratory reference ranges: ALT or AST level > 5 times the upper limit of normal (ULN) OR ALT or AST > 3 times the ULN and total bilirubin level > 2 times the ULN
* Pregnant or breastfeeding, or positive pregnancy test in a predose examination, or intending to become pregnant during the study or within 28 days after the last dose of study treatment
* Exposure to an investigational drug within 5 half-lives or 30 days (whichever is longer) of randomization
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study
* Known hypersensitivity to baloxavir marboxil or the drug product excipients
* Known COVID-19 coinfection
* Unwilling to undergo nasopharyngeal (NP) swabs as per study schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mirella Salvatore, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burnham P, Khush K, De Vlaminck I. Myriad Applications of Circulating Cell-Free DNA in Precision Organ Transplant Monitoring. Ann Am Thorac Soc. 2017 Sep;14(Supplement_3):S237-S241. doi: 10.1513/AnnalsATS.201608-634MG. PMID 28945480
- [Background] de Jong MD, Ison MG, Monto AS, Metev H, Clark C, O'Neil B, Elder J, McCullough A, Collis P, Sheridan WP. Evaluation of intravenous peramivir for treatment of influenza in hospitalized patients. Clin Infect Dis. 2014 Dec 15;59(12):e172-85. doi: 10.1093/cid/ciu632. Epub 2014 Aug 12. PMID 25115871
- [Background] De Vlaminck I, Martin L, Kertesz M, Patel K, Kowarsky M, Strehl C, Cohen G, Luikart H, Neff NF, Okamoto J, Nicolls MR, Cornfield D, Weill D, Valantine H, Khush KK, Quake SR. Noninvasive monitoring of infection and rejection after lung transplantation. Proc Natl Acad Sci U S A. 2015 Oct 27;112(43):13336-41. doi: 10.1073/pnas.1517494112. Epub 2015 Oct 12. PMID 26460048
- [Background] De Vlaminck I, Valantine HA, Snyder TM, Strehl C, Cohen G, Luikart H, Neff NF, Okamoto J, Bernstein D, Weisshaar D, Quake SR, Khush KK. Circulating cell-free DNA enables noninvasive diagnosis of heart transplant rejection. Sci Transl Med. 2014 Jun 18;6(241):241ra77. doi: 10.1126/scitranslmed.3007803. PMID 24944192
- [Background] Fiore AE, Fry A, Shay D, Gubareva L, Bresee JS, Uyeki TM; Centers for Disease Control and Prevention (CDC). Antiviral agents for the treatment and chemoprophylaxis of influenza --- recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Recomm Rep. 2011 Jan 21;60(1):1-24. PMID 21248682
- [Background] Fukao K, Ando Y, Noshi T, Kitano M, Noda T, Kawai M, Yoshida R, Sato A, Shishido T, Naito A. Baloxavir marboxil, a novel cap-dependent endonuclease inhibitor potently suppresses influenza virus replication and represents therapeutic effects in both immunocompetent and immunocompromised mouse models. PLoS One. 2019 May 20;14(5):e0217307. doi: 10.1371/journal.pone.0217307. eCollection 2019. PMID 31107922
- [Background] Fukao K, Noshi T, Yamamoto A, Kitano M, Ando Y, Noda T, Baba K, Matsumoto K, Higuchi N, Ikeda M, Shishido T, Naito A. Combination treatment with the cap-dependent endonuclease inhibitor baloxavir marboxil and a neuraminidase inhibitor in a mouse model of influenza A virus infection. J Antimicrob Chemother. 2019 Mar 1;74(3):654-662. doi: 10.1093/jac/dky462. PMID 30476172
- [Background] Hayden FG, Sugaya N, Hirotsu N, Lee N, de Jong MD, Hurt AC, Ishida T, Sekino H, Yamada K, Portsmouth S, Kawaguchi K, Shishido T, Arai M, Tsuchiya K, Uehara T, Watanabe A; Baloxavir Marboxil Investigators Group. Baloxavir Marboxil for Uncomplicated Influenza in Adults and Adolescents. N Engl J Med. 2018 Sep 6;379(10):913-923. doi: 10.1056/NEJMoa1716197. PMID 30184455
- [Background] Harper SA, Bradley JS, Englund JA, File TM, Gravenstein S, Hayden FG, McGeer AJ, Neuzil KM, Pavia AT, Tapper ML, Uyeki TM, Zimmerman RK; Expert Panel of the Infectious Diseases Society of America. Seasonal influenza in adults and children--diagnosis, treatment, chemoprophylaxis, and institutional outbreak management: clinical practice guidelines of the Infectious Diseases Society of America. Clin Infect Dis. 2009 Apr 15;48(8):1003-32. doi: 10.1086/598513. PMID 19281331
- [Background] Hu Y, Lu S, Song Z, Wang W, Hao P, Li J, Zhang X, Yen HL, Shi B, Li T, Guan W, Xu L, Liu Y, Wang S, Zhang X, Tian D, Zhu Z, He J, Huang K, Chen H, Zheng L, Li X, Ping J, Kang B, Xi X, Zha L, Li Y, Zhang Z, Peiris M, Yuan Z. Association between adverse clinical outcome in human disease caused by novel influenza A H7N9 virus and sustained viral shedding and emergence of antiviral resistance. Lancet. 2013 Jun 29;381(9885):2273-9. doi: 10.1016/S0140-6736(13)61125-3. Epub 2013 May 29. PMID 23726392
- [Background] Lee N, Chan PK, Hui DS, Rainer TH, Wong E, Choi KW, Lui GC, Wong BC, Wong RY, Lam WY, Chu IM, Lai RW, Cockram CS, Sung JJ. Viral loads and duration of viral shedding in adult patients hospitalized with influenza. J Infect Dis. 2009 Aug 15;200(4):492-500. doi: 10.1086/600383. PMID 19591575
- [Background] Lee N, Ison MG. Diagnosis, management and outcomes of adults hospitalized with influenza. Antivir Ther. 2012;17(1 Pt B):143-57. doi: 10.3851/IMP2059. Epub 2012 Feb 3. PMID 22311561
- [Background] Marty FM, Vidal-Puigserver J, Clark C, Gupta SK, Merino E, Garot D, Chapman MJ, Jacobs F, Rodriguez-Noriega E, Husa P, Shortino D, Watson HA, Yates PJ, Peppercorn AF. Intravenous zanamivir or oral oseltamivir for hospitalised patients with influenza: an international, randomised, double-blind, double-dummy, phase 3 trial. Lancet Respir Med. 2017 Feb;5(2):135-146. doi: 10.1016/S2213-2600(16)30435-0. Epub 2017 Jan 14. PMID 28094141
- [Background] Muthuri SG, Venkatesan S, Myles PR, Leonardi-Bee J, Al Khuwaitir TS, Al Mamun A, Anovadiya AP, Azziz-Baumgartner E, Baez C, Bassetti M, Beovic B, Bertisch B, Bonmarin I, Booy R, Borja-Aburto VH, Burgmann H, Cao B, Carratala J, Denholm JT, Dominguez SR, Duarte PA, Dubnov-Raz G, Echavarria M, Fanella S, Gao Z, Gerardin P, Giannella M, Gubbels S, Herberg J, Iglesias AL, Hoger PH, Hu X, Islam QT, Jimenez MF, Kandeel A, Keijzers G, Khalili H, Knight M, Kudo K, Kusznierz G, Kuzman I, Kwan AM, Amine IL, Langenegger E, Lankarani KB, Leo YS, Linko R, Liu P, Madanat F, Mayo-Montero E, McGeer A, Memish Z, Metan G, Mickiene A, Mikic D, Mohn KG, Moradi A, Nymadawa P, Oliva ME, Ozkan M, Parekh D, Paul M, Polack FP, Rath BA, Rodriguez AH, Sarrouf EB, Seale AC, Sertogullarindan B, Siqueira MM, Skret-Magierlo J, Stephan F, Talarek E, Tang JW, To KK, Torres A, Torun SH, Tran D, Uyeki TM, Van Zwol A, Vaudry W, Vidmar T, Yokota RT, Zarogoulidis P; PRIDE Consortium Investigators; Nguyen-Van-Tam JS. Effectiveness of neuraminidase inhibitors in reducing mortality in patients admitted to hospital with influenza A H1N1pdm09 virus infection: a meta-analysis of individual participant data. Lancet Respir Med. 2014 May;2(5):395-404. doi: 10.1016/S2213-2600(14)70041-4. Epub 2014 Mar 19. PMID 24815805
- [Background] Paules C, Subbarao K. Influenza. Lancet. 2017 Aug 12;390(10095):697-708. doi: 10.1016/S0140-6736(17)30129-0. Epub 2017 Mar 13. PMID 28302313
- [Background] Rothberg MB, Haessler SD. Complications of seasonal and pandemic influenza. Crit Care Med. 2010 Apr;38(4 Suppl):e91-7. doi: 10.1097/CCM.0b013e3181c92eeb. PMID 19935413
- [Background] Salvatore M, Laplante JM, Soave R, Orfali N, Plate M, van Besien K, St George K. Baloxavir for the treatment of Influenza in allogeneic hematopoietic stem cell transplant recipients previously treated with oseltamivir. Transpl Infect Dis. 2020 Aug;22(4):e13336. doi: 10.1111/tid.13336. Epub 2020 Jun 10. PMID 32449254
- [Background] Taniguchi K, Ando Y, Nobori H, Toba S, Noshi T, Kobayashi M, Kawai M, Yoshida R, Sato A, Shishido T, Naito A, Matsuno K, Okamatsu M, Sakoda Y, Kida H. Inhibition of avian-origin influenza A(H7N9) virus by the novel cap-dependent endonuclease inhibitor baloxavir marboxil. Sci Rep. 2019 Mar 5;9(1):3466. doi: 10.1038/s41598-019-39683-4. PMID 30837531
- See also: Influenza Antiviral Medications: Summary for Clinicians — https://www.cdc.gov/flu/hcp/antivirals/summary-clinicians.html?CDC_AAref_Val=https://www.cdc.gov/flu/professionals/antivirals/summary-clinicians.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study was challenging because of changed flu seasonality and low flu cases following covid-19
Period: Overall Study
Arm/Group | Active and Standard of Care | Placebo and Standard of Care
Started | 0 | 2
Completed | 0 | 1
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants were not analyzed in the Active and Standard of Care arm because 0 participants were enrolled in that arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active and Standard of Care | Placebo and Standard of Care | Total
Number analyzed (Participants) | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 45 (30) | 45 (30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 1 | 1
  Not Hispanic or Latino |  | 1 | 1
  Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 1 | 1
  White |  | 1 | 1
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change of Influenza Viral RNA Loads From Baseline at the End of Treatment as Measured by Quantitative Real Time Polymerase Chain Reaction.
Description: Influenza viral RNA loads will be measured by quantitative real time polymerase chain reaction.
Time Frame: Baseline; Day 10
Population: The only patient that completed the study, was randomized into the placebo arm.
Measure: Number; unit: copies per mL
Arm/Group | Active and Standard of Care | Placebo and Standard of Care
Number analyzed (Participants) | 0 | 1
copies per mL
  Baseline |  | 2300000
  Day 10 |  | 0

2. Primary Outcome: Between-treatment-arm Difference in the Change of Influenza Viral RNA Loads From Baseline at the End of Treatment as Measured by Quantitative Real Time Polymerase Chain Reaction.
Description: Influenza viral load will be measured by the quantitative real time polymerase chain reaction.
Time Frame: Baseline; Day 10
Population: The only patient that completed the study, was randomized into the placebo arm. Difference cannot be calculated as one arm has zero patients.
Measure: Number; unit: copies per mL
Arm/Group | Active and Standard of Care | Placebo and Standard of Care
Number analyzed (Participants) | 0 | 1
copies per mL
  Baseline |  | 2300000
  Day 10 |  | 0

3. Primary Outcome: Between-treatment-arm Difference in the Change of Influenza Viral RNA Loads From Baseline at the End of Treatment as Measured by Influenza Plaque Assay (Replicating Virus).
Description: Influenza viral load will be measured by the influenza plaque assay.
Time Frame: Baseline; Day 10
Population: as for outcome 2
Measure: Number; unit: PFU per mL
Arm/Group | Active and Standard of Care | Placebo and Standard of Care
Number analyzed (Participants) | 0 | 1
PFU per mL
  Baseline |  | 2300000
  Day 10 |  | 0

4. Secondary Outcome: Change of Influenza Viral RNA Load From Baseline at Day 4 and Day 7 and 10 in Each Treatment Arm
Description: Influenza viral RNA load will be measured by quantitative real time polymerase chain reaction.
Time Frame: Baseline; Day 4; Day 7; Day 10
Population: The only patient that completed the study, was randomized into the placebo arm.
Measure: Number; unit: copies per mL
Arm/Group | Active and Standard of Care | Placebo and Standard of Care
Number analyzed (Participants) | 0 | 1
copies per mL
  Baseline |  | 2300000
  Day 4 |  | 800
  Day 7 |  | 1300
  Day 10 |  | 0

5. Secondary Outcome: Difference in Change of Influenza Viral Loads From Baseline at Day 4, 7 and 10 Between the Two Treatment Arms as Measured by Quantitative Real Time Polymerase Chain Reaction
Description: Influenza viral RNA load will be measured by quantitative real time polymerase chain reaction.
Time Frame: Baseline; Day 4; Day 7; Day 10
Population: as for outcome 2
Measure: Number; unit: copies per mL
Arm/Group | Active and Standard of Care | Placebo and Standard of Care
Number analyzed (Participants) | 0 | 1
copies per mL
  Baseline |  | 2300000
  Day 4 |  | 800
  Day 7 |  | 1300
  Day 10 |  | 0

6. Secondary Outcome: Change of Influenza Viral Loads From Baseline at Day 4, 7 and 10 as Measured by Influenza Plaque Assay (Replicating Virus) in Each Treatment Arm
Description: Influenza viral load will be measured by the influenza plaque assay (replicating virus).
Time Frame: Baseline; Day 4; Day 7; Day 10
Population: The only patient that completed the study, was randomized into the placebo arm.
Measure: Number; unit: PFU per mL
Arm/Group | Active and Standard of Care | Placebo and Standard of Care
Number analyzed (Participants) | 0 | 1
PFU per mL
  Baseline |  | 2300000
  Day 4 |  | 800
  Day 7 |  | 1300
  Day 10 |  | 0

7. Secondary Outcome: Difference in Change of Influenza Viral Loads From Baseline at Day 4, 7 and 10 Between the Two Treatment Arms as Measured by Influenza Plaque Assay (Replicating Virus)
Description: Influenza viral load will be measured by the influenza plaque assay (replicating virus).
Time Frame: Baseline; Day 4; Day 7; Day 10
Population: as for outcome 2
Measure: Number; unit: PFU per mL
Arm/Group | Active and Standard of Care | Placebo and Standard of Care
Number analyzed (Participants) | 0 | 1
PFU per mL
  Baseline |  | 2300000
  Day 4 |  | 800
  Day 7 |  | 1300
  Day 10 |  | 0

8. Secondary Outcome: Time to Improvement of Individual Influenza Symptoms as Assessed by Patient-reported Outcome Measures on a Single Scale
Description: Patients will self-assess the severity of 7 influenza-associated symptoms on a 4-point single scale with 0 indicating no symptoms and higher scores indicating mild, moderate, and severe symptoms. Time to improvement of individual influenza symptoms are defined as the time from the start of treatment to the time when each of the influenza symptoms are alleviated, maintained, or improved for a duration of at least 21.5 hours. These are defined as: pre-existing symptoms (cough, fatigue, or muscle/join pain that existed prior to influenza) that were worse at baseline and had improved at least 1 point from baseline; pre-existing symptoms not worse at baseline that maintained baseline severity; and new symptoms that were alleviated, defined as a symptom score of non (0) or mild (1).
Time Frame: Baseline to Day 30
Population: The only patient that completed the study, was randomized into the placebo arm.
Measure: Number; unit: Days to recovery
Arm/Group | Active and Standard of Care | Placebo and Standard of Care
Number analyzed (Participants) | 0 | 1
Days to recovery |  | 8

9. Secondary Outcome: Percentage of Patients Who Experience Each Influenza-related Complications: Hospitalization, Death, Sinusitis, Otitis Media, Bronchitis, and Radiologically-confirmed Pneumonia as an Adverse Event After the Initiation of Study Treatment
Description: A composite score of multiple measures will be used and calculated by count of patients who experience each influenza-related complications. Adverse events will only include those that are determined to be related to the study drug.
Time Frame: Day 1 to Day 30
Population: The only patient that completed the study, was randomized into the placebo arm.
Measure: Number; unit: Number of patients with complications.
Arm/Group | Active and Standard of Care | Placebo and Standard of Care
Number analyzed (Participants) | 0 | 1
Number of patients with complications. |  | 0

10. Secondary Outcome: Time to Return to Preinfluenza Health Status
Description: Preinfluenza health status will be measured on a score from 0 (worst possible health) to 10 (normal health [for someone your age and condition]).
Time Frame: Day 1 to Day 30
Population: The only patient that completed the study, was randomized into the placebo arm.
Measure: Number; unit: Days
Arm/Group | Active and Standard of Care | Placebo and Standard of Care
Number analyzed (Participants) | 0 | 1
Days |  | 8

11. Secondary Outcome: Time to Viral Clearance, as Assessed by Difference in Percentage of Participants Positive by Influenza Plaque Assay at Each Time-point (in Each Treatment Group)
Description: Time to viral clearance will be assessed by percentage of participants positive by influenza plaque assay at each time-point.
Time Frame: Baseline to Day 30
Population: The only patient that completed the study, was randomized into the placebo arm.
Measure: Number; unit: Days
Arm/Group | Active and Standard of Care | Placebo and Standard of Care
Number analyzed (Participants) | 0 | 1
Days |  | 8

12. Secondary Outcome: Time to Viral Clearance, as Assessed by Difference in Percentage of Participants Positive by Quantitative Real Time Polymerase Chain Reaction
Description: Time to viral clearance will be assessed by percentage of participants positive by qPCR at each time-point.
Time Frame: Baseline to Day 30
Population: The only patient that completed the study, was randomized into the placebo arm.
Measure: Number; unit: Days
Arm/Group | Active and Standard of Care | Placebo and Standard of Care
Number analyzed (Participants) | 0 | 1
Days |  | 8

13. Secondary Outcome: Change of Treatment-emergent Variants of Neuraminidase and Polymerase Known to Confer Antiviral Resistance to Oseltamivir in Each Arm by Direct Next-generation Sequencing Symptoms
Description: Treatment-emergent variants will be identified using direct next-generation sequencing of a comprehensive panel of genes.
Time Frame: Baseline to Day 30
Population: The only patient that completed the study, was randomized into the placebo arm.
Measure: Number; unit: Resistant variant
Arm/Group | Active and Standard of Care | Placebo and Standard of Care
Number analyzed (Participants) | 0 | 1
Resistant variant |  | 0

14. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: Adverse events will only include those that are determined to be related to the study drug and will assess the safety and tolerability of Baloxavir in Combination with SOC treatment.
Time Frame: Day 1 to Day 15
Population: The only patient that completed the study, was randomized into the placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Active and Standard of Care | Placebo and Standard of Care
Number analyzed (Participants) | 0 | 1
Participants |  | 1

ADVERSE EVENTS:
Time Frame: 1 month
Description: 0 Participants were analyzed in the Active and Standard of Care arm because 0 subjects were enrolled in that arm.
Arm/Group | Active and Standard of Care | Placebo and Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 1/2
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/2
Other Adverse Events (participants affected / at risk) | 0/0 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active and Standard of Care (N=0) | Placebo and Standard of Care (N=2)
renal insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1) — Participant developed renal failure independently from study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active and Standard of Care (N=0) | Placebo and Standard of Care (N=2)
alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Participant stated that she noticed increased hair loss during treatment

LIMITATIONS AND CAVEATS:
Due to change in patterns of respiratory viruses, and low or no flu circulating, we were unable to enroll the target number of participants. The only participants enrolled were the 2 in the placebo arm, 1 of whom withdrew early on. No comparison is possible with only 1 placebo participant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-05): https://cdn.clinicaltrials.gov/large-docs/09/NCT05170009/Prot_SAP_000.pdf